CLINICAL TRIAL: NCT04255108
Title: Validation of a Sensor for Non-invasive Measurement of Stroke Volume and Cardiac Output
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: TS-IRB-0003.1
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Cardiac Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Men/Women who meet the inclusion/exclusion criteria
  Interventions: Device: Cova Patch

INTERVENTIONS:
Device: Cova Patch — CoVa Patch will measure quasi-continuously, approximately every 5 minutes for a period between 6 to 48 hours

SUMMARY:
toSense, Inc. has developed a novel, non-invasive, body-worn sensor -CoVa Patch-that offers an alternative to invasive continuous cardiac output monitoring. To validate this new sensor's measurements of stroke volume and cardiac output, toSense, Inc. will conduct a study that compares its measurement performance to that from a pulmonary artery catheter using the thermodilution method.

DETAILED DESCRIPTION:
This in an introductory clinical study with cardiac ICU patients featuring CoVa Patch. This is a single site, non-blinded, non-randomized study. It will employ a retrospective analysis comparing the accuracy of SV and CO. The 'test sensor', CoVa Patch, which will measure SV and CO quasi-continuously and non-invasively, approximately every 5-30 minutes for a period of time lasting approximately 12-48 hours. These measurements will be compared to those from a 'reference device', which is the pulmonary arterial catheter. It uses an invasive technique called thermodilution that will be made approximately every 4 hours. Measurements between the test and reference devices will be compared in a retrospective analysis once the study has completed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at Visit X.
* Subject is a patient in the Cardiac ICU and meets the following criteria: pulmonary artery catheterization scheduled or completed.
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
* Subject is not pregnant at the time of consent

Exclusion Criteria:

* Pregnant in the study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Subject is unable or unwilling to wear electrode patches as required for a period between 6 to 48 hours.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men and woman over the age of 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Accuracy of Stroke Volume | 4 Months
  The primary objective of this study is to validate stroke volume (the amount of blood pumped by the left ventrical of the heart in one contraction) measurements made using CoVa Patch to those made using a pulmonary artery catheter and the thermodilution method.
  Thermodilution requires a pulmonary artery catheter and are calculated by a monitoring system based on temperature changes in the heart when a cooler solution is injected into the right atrium via the proximal port of a pulmonary artery catheter.
Accuracy of Cardiac Output | 4 Months
  The secondary objective of this study is to validate cardiac output (the amount of blood the heart pumps per minute) measurements made using CoVa Patch to those made using a pulmonary artery catheter and the thermodilution method.
  Thermodilution requires a pulmonary artery catheter and are calculated by a monitoring system based on temperature changes in the heart when a cooler solution is injected into the right atrium via the proximal port of a pulmonary artery catheter.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiac ICU, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No